CLINICAL TRIAL: NCT05958056
Title: The Acute Effect of Low Load Resistance Exercises With Blood Flow Restriction Versus High Load Resistance Exercises on Growth Hormone and Blood Lactate
Brief Title: Low Load Resistance Exercises With Blood Flow Restriction Versus High Load Resistance Exercises
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jordan (Other)
Collaborators: The Hashemite University (Other)
Responsible Party: Principal Investigator, Alia A. Alghwiri, Professor, University of Jordan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 4/2019
Record Dates: First submitted 2023-07-14; First posted 2023-07-24 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Athletes
Keywords: blood flow restriction; Growth hormone; Blood lactate
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low load resistance exercises with Practical blood flow restriction (PBFR) (Experimental): Participants in the experimental group performed one session of 30% 1RM with Practical blood flow restriction training. The number of repetitions in every set was 15 times with PBFR.19 Participants in the experimental group used the elite band (occlusion training bands) for both thighs during the training session. The width of the thigh band was 5cm, which would produce a pressure between 160-240 mmHg. This pressure range is appropriate for most of the individuals who used PBFR.27 The perceived pressure scale (PPS) was used to estimate the appropriate pressure (7 out of 10) in training before performing the exercises.28,29 The blood flow restriction bands booklet was used30 along with previous studies to design the training session. Participants removed the BFR band immediately after the end of the training session.
  Interventions: Other: Resistance exercise
- High resistance exercises (Active Comparator): Participants in the control group performed one session of 80% 1RM without PBFR. The number of repetitions in every set was 10 times.
  Interventions: Other: Resistance exercise

INTERVENTIONS:
Other: Resistance exercise — The training session included leg curl and leg extension exercises with 4 sets each. Participants started with leg extension exercise for 4 sets with a 30-second rest periods between the sets. Then, participants took a rest for 60 seconds. Afterward, participants performed leg curl exercise for 4 sets with a 30-second rest periods between the sets. Exercises in each set were performed continuously (uninterrupted) with a speed of 2 seconds for each repetition and a medium exercise performance speed.

SUMMARY:
Practical blood flow restriction (PBFR) is a new technique of reducing the venous return using a band with a pressure that is applied using a perceived pressure scale. The studies that investigate the acute effect of using PBFR and regular high intensity exercises on the level of growth hormone (GH) and blood lactate (BL) after lower extremity training in collegiate athletes are scarce.

DETAILED DESCRIPTION:
Practical blood flow restriction (PBFR) is a new technique of reducing the venous return using a band with a pressure that is applied using a perceived pressure scale. The studies that investigate the acute effect of using PBFR and regular high intensity exercises on the level of growth hormone (GH) and blood lactate (BL) after lower extremity training in collegiate athletes are scarce. Therefore, this study aimed to investigate the acute effect of a single session low load resistance exercises with PBFR compared to a high load resistance exercises without PBFR on the levels of GH and BL. A convenience sample of collegiate athletes were allocated to either an experimental group that performed low resistance exercises with PBFR or a control group that performed high resistance exercises without PBFR. The levels of GH and BL were examined in 3 time points: pre-training, immediate post-training, and 15 minutes post-training for both groups. Analysis of Variance (ANOVA) was used to assess the main and interaction effects of the groups.

ELIGIBILITY:
Inclusion Criteria:

* Student collegiate athletes.
* Age of 18 years and older.
* Free from any cardiovascular or respiratory disorders and did not have any injuries during the previous 12 months.

Exclusion Criteria:

* Students who were taking any medications for chronic conditions.
* Student who were taking any supplements.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Growth Hormone | Before intervention.
  Blood test of the level of growth hormone
Growth Hormone | Immediately post intervention.
  Blood test of the level of growth hormone
Growth Hormone | 15 minutes after the end of intervention.
  Blood test of the level of growth hormone
Blood lactate | Before intervention.
  Blood test of the level of Blood lactate
Blood lactate | Immediately post intervention.
  Blood test of the level of Blood lactate
Blood lactate | 15 minutes after the end of intervention.
  Blood test of the level of Blood lactate

CONTACTS AND LOCATIONS:
Overall Officials: Alia Alghwiri, PhD, Study Director — The University of Jordan
Locations (1):
- The University of Jordan, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No